CLINICAL TRIAL: NCT01591343
Title: Prospective Study to Evaluate the Safety of a 4-month Treatment With Depigoid® Dermatophagoides Pteronyssinus or 50% Dermatophagoides Pteronyssinus / 50% Dermatophagoides Farinae (500 DPP/ml) in Patients With Allergic Rhinitis or Rhinoconjunctivitis With or Without Mild Persistent or Intermittent Asthma
Brief Title: Safety Study of Depigoid Vaccine Dermatophagoides Pteronyssinus or 50% Dermatophagoides Pteronyssinus / 50% Dermatophagoides Farinae (500 DPP/ml), to Treat Allergic Rhinitis or Rhinoconjunctivitis With or Without Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted by Sponsor
Sponsor: Laboratorios Leti, S.L. (Industry)
Collaborators: Harrison Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 101-PG-PSC-186
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Allergic Rhinitis; Rhinoconjunctivitis; Mild Persistent Asthma; Mild Intermittent Asthma
Keywords: Specific immunotherapy; Allergic rhinitis; Allergic rhinoconjunctivitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Depigoid® (500 DPP/ml) (Experimental): Patients will receive either Depigoid® Dermatophagoides pteronyssinus or 50% Dermatophagoides pteronyssinus / 50% Dermatophagoides farinae (500 DPP/ml), depending on their sensitization to one or both mites (Dermatophagoides pteronyssinus and Dermatophagoides farinae).
  Interventions: Biological: Depigoid® (500 DPP/ml)

INTERVENTIONS:
Biological: Depigoid® (500 DPP/ml) — Depigoid® D. pteronyssinus or Depigoid® 50% D. pteronyssinus / 50% D. farinae (500 DPP/ml).
  Dose:
  Week 0: 0.2 ml followed by 0.3 ml after 30 min Week 4, 8, 12, and 16: 0.5 ml Mode of administration: subcutaneous injection

SUMMARY:
Safety study of Depigoid vaccine Dermatophagoides pteronyssinus or 50% Dermatophagoides pteronyssinus / 50% Dermatophagoides farinae (500 DPP/ml), to treat allergic rhinitis or rhinoconjunctivitis with or without asthma.

Primary variable: number of subjects [%] who experienced at least one immediate or delayed systemic reaction of EAACI grade 2 or higher during the 4-month treatment period.

DETAILED DESCRIPTION:
Investigator(s):

Approximately 10 study centers (allergy services) in Spain

Planned study period:

MAY 2012 (first subject in) - MAR 2013 (last subject out)

Objectives:

Primary objective: to evaluate the safety of a 4-month treatment with an extract of Depigoid® Dermatophagoides pteronyssinus or a mixture of 50% Dermatophagoides pteronyssinus and 50% Dermatophagoides farinae at a concentration of 500 DPP/ml administered following a rush build-up regimen.

Secondary objective: to assess the subjects' immunologic responses to the above treatment.

Study design:

This is a prospective, non-randomized, uncontrolled, open-label safety study. When the first 29 subjects have completed the study, an interim analysis will be conducted to check whether the number of systemic reactions in these subjects is below a predefined limit.

Planned number of subjects:

103 subjects in total.

Medical condition or disease under investigation:

Allergic rhinitis or rhinoconjunctivitis, with or without mild persistent or intermittent asthma.

Test product, dose and mode of administration:

Depigoid® D. pteronyssinus or Depigoid® 50% D. pteronyssinus / 50% D. farinae (500 DPP/ml).

Dose: Week 0: 0.2 ml followed by 0.3 ml after 30 min Week 4, 8, 12, and 16: 0.5 ml Mode of administration: subcutaneous injection

Duration of treatment:

16 weeks.

Criteria for evaluation:

Safety:

Local and systemic adverse reactions (EAACI classification); adverse events.

Efficacy:

Immunologic response to the treatment.

Statistical methods:

Primary variable: number of subjects [%] who experienced at least one immediate or delayed systemic reaction of EAACI grade 2 or higher during the 4-month treatment period.

Analysis of primary variable: exact binomial test

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 55 years of age (both inclusive).
* Individuals suffering symptoms of allergic rhinoconjunctivitis or rhinitis during at least the preceding year -- with or without symptoms of mild persistent or intermittent allergic asthma which is controlled with a dose less or equal to 400 µg/day budesonide or an equivalent -- caused by a clinically relevant sensitization to house dust mites (Dermatophagoides pteronyssinus or Dermatophagoides pteronyssinus and Dermatophagoides farinae).
* The IgE-mediated sensitization will be demonstrated by means of the following: medical history and IgE specific to house dust mites (D. pteronyssinus or D. pteronyssinus and D. farinae) CAP RAST ≥ 2 and positive skin prick test. A skin prick test will be considered positive when it produces a wheal of at least 3 mm according to the largest diameter.
* Asthmatic patients must be stable and on a stable inhaled steroid dose within 6 weeks prior to visit 1 and throughout the study.

Exclusion Criteria:

* Any contraindication for treatment with allergen specific immunotherapy.
* Forced expiratory volume in 1 s (FEV1) or peak expiratory flow (PEF) value < 80% of the predicted normal value.
* Allergy symptoms due to sensitization to pollens or other perennial allergens (molds, epithelia).
* Subjects with typical symptoms to co-allergens such as tree pollen, grasses or weeds, fungi or animal epithelial cells cannot participate in this study. Patients sensitized to pollens with specific IgE CAP RAST < 2 can be included in this study provided that they do not present symptoms as a consequence of this sensitization. Patients sensitized to animal epithelia who do not present symptoms can participate in this study provided that they are not exposed to the allergen to which they are sensitized, even though they present specific IgE with CAP RAST ≥ 2. If they were exposed to the animal in question, these subjects must have a specific IgE with CAP RAST < 2 in order to participate in the study.
* Asthma requiring a dose > 400 µg/day of Budesonide or an equivalent, without long-lasting beta-2 agonists, to reach control according to the Global Initiative for Asthma (GINA 2010).
* Patients with non controlled bronchial asthma within 3 months prior to Visit 1.
* Patients with asthma who have been treated with systemic steroids within 3 months prior to V1.
* Patients with hospital admission due to asthma exacerbations within 1 year prior to V1
* Acute or chronic inflammatory or infectious diseases of the airways.
* Chronic structural diseases of the respiratory system (for example, emphysema or bronchiectasis).
* Immune system diseases, both autoimmune diseases and immunodeficiency.
* Any disease involving a contraindication for the use of adrenaline (for example, hyperthyroidism).
* Serious uncontrolled diseases involving a risk for the subjects participating in this study, including the following for example: heart failure, serious or uncontrolled respiratory diseases, endocrine diseases, clinically relevant liver or kidney diseases or hematological diseases.
* Malignant disease with activity in the last 5 years.
* Clinically significant anomaly in laboratory parameters or vital signs which could involve a risk increase for the subject.
* Excessive consumption of alcohol, drugs or medication in the preceding year.
* Serious psychiatric, psychological or neurological disorders.
* Use of immunotherapy with allergenic extracts of storage or house dust mites in the last 5 years.
* Systemic or topical treatment with beta-blocker drugs.
* Treatment with substances interfering with the immune system 2 weeks before visit 2.
* Use of psychotropic or antidepressants substances.
* Use of systemic corticosteroids 3 months before visit 1.
* Immunization with prophylactic (bacterial or viral) vaccines within 7 days before visit 2. (Prophylactic vaccines are allowed during the administration of IMP period provided they are administered at least one week after immunotherapy and the next immunotherapy dose is administered at least 14 days later).
* Participation of the subject in another clinical trial 30 days before visit 2.
* Subjects who have already participated in this clinical trial.
* Subjects who are going to donate stem cells, blood, organs or bone marrow in the course of the study.
* Female subjects who are pregnant or nursing and women with a positive pregnancy test at visit 1 or 2.
* Women of childbearing potential not using highly effective methods of birth control. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomized partner. Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.
* No written informed consent upon enrolment.
* Not willing to give consent for transmission of personal "pseudonymised" data.
* Subjects who are unable to comply with the requirements of the study or who in the opinion of the investigator should not participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Primary variable | 4 months
  Number of subjects [%] who experienced at least one immediate or delayed systemic reaction of EAACI grade 2 or higher during the 4-month treatment period.

SECONDARY OUTCOMES:
Secondary variables | 4 months
  Secondary variables, which will be analyzed descriptively, are the
  * Number of subjects [%] suffering immediate and/or delayed systemic reactions broken down by grade (EAACI classification).
  * Number of subjects [%] suffering immediate and/or delayed local reactions broken down by diameter (< 5 cm, 5-10 cm or > 10 cm).
  * Number of immediate and/or delayed systemic reactions broken down by grade (EAACI classification).
  * Number of immediate and/or or delayed local reactions broken down by diameter (< 5 cm, 5-10 cm and > 10 cm).
  * Immunologic response to the treatment.

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Complejo Hospitalario Torrecárdenas, Almería, Andalusia
  - Clínica Doctor Lobatón, Cadiz, Andalusia
  - Hospita Universitario Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Al·lergo Centre, Barcelona, Catalonia
  - Centro Médico Teknon, Barcelona, Catalonia
  - Hospital Universitario Vall d'Hebrón, Barcelona, Catalonia
  - Hospital Universitario de Bellvitge, Barcelona, Catalonia
  - Hospital Universitario Joan XXIII, Tarragona, Catalonia
  - Complejo Hospitalario Universitario de Cartagena, Cartagena, Murcia